CLINICAL TRIAL: NCT04053647
Title: Quality of Life Evaluation (SF-36) in Patients With Permanent Hypoparathyroidism After Total Thyroidectomy
Brief Title: Quality of Life Evaluation (SF-36) in Patients With Permanent Hypoparathyroidism After Total Thyroidectomy (Qol-Hypopara)
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: University Hospital, Angers (Other Government); Centre Hospitalier le Mans (Other); University Hospital, Limoges (Other); Central Hospital, Nancy, France (Other); Pitié-Salpêtrière Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC19_0021
Record Dates: First submitted 2019-05-22; First posted 2019-08-12 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Hypoparathyroidism; Quality of Life
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypoparathyroid patients: Patients with persistent hypoparathyroidism after total thyroidectomy, defined as serum PTH inferior to 15 pg/mL 6 months after surgery and the need of vitamin-calcic supplementation.
  Interventions: Other: Non-interventional study
- Control patients, without hypoparathyroidism
  Interventions: Other: Non-interventional study

INTERVENTIONS:
Other: Non-interventional study — Non-interventional study

SUMMARY:
Persistent hypoparathyroidism is an underestimate but major complication of total thyroidectomy. The hypothesis of the investigators is that the mental health is impaired in hypoparathyroid patients compared with thyroidectomized patients without hypoparathyroidism. The investigators evaluated the quality of life using the SF-36 survey in comparison with a control population of patients thyroidectomized but free from this complication. The voice quality, the cardiovascular risk, the kidney function and the incidence of urinary lithiasis were also evaluated.

DETAILED DESCRIPTION:
Persistent hypoparathyroidism is an underestimate but major complication of total thyroidectomy. In this retrospective, observational, multicentre study, the investigators evaluated the quality of life using the SF-36 survey in comparison with a control population of patients thyroidectomized but free from this complication. Patients in six centers in France (Angers, Le Mans, Limoges, Nancy, Nantes, la Pitié-Salpétrière) and in the association "Hypoparathyroïdisme France" were contacted by mail. The primary endpoint was the mental health. The physic and global quality of life scores were assessed as secondary endpoints. Medical and VHI surveys were also send to the patients. The voice quality, the cardiovascular risk, the kidney function and the incidence of urinary lithiasis were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated of total thyroidectomy
* Patients suffering from persistent hypoparathyroidism defined as serum PTH inferior to 15 pg/mL 6 months after the surgery, requiring vitamin-calcic supplementation.
* Age superior to 18
* Answering the survey

Exclusion Criteria:

* Pregnancy at the time of the study
* Age inferior to 18 or adult under guardianship
* Patients with vitamino-calcic supplementation without serum PTH measurement
* Cause of hypoparathyroidism other than post-operatory.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is that of hypoparathyroid patients of the Hypoparathyroidism France combination who have undergone total thyroidectomy and who have agreed to participate in the study.
  Patients with permanent hypoparathyroidism who were included in the ThyrQol study and in the FOTHYR study will also be solicited. Endocrinologists at the University Hospital of Nantes also have patients with permanent hypoparathyroidism in their patients.
  The control population consists of patients who had a total thyroidectomy and were included in the ThyrQol study between 2014 and 2018, without sequelary hypoparathyroidism.
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Mental health | Through study completion, an average of 1 year
  Items from mental quality of life score defined by the SF36 (Short Form 36) survey

SECONDARY OUTCOMES:
Physical quality score | Through study completion, an average of 1 year
  Items from the SF36 (Short Form 36) survey
Global quality of life score | Through study completion, an average of 1 year
  Items from the SF36 (Short Form 36) survey
Voice quality | Through study completion, an average of 1 year
  Items from the VHI (Voice Handicap Index) survey
Renal function quality | Through study completion, an average of 1 year
  Serum creatinine and clearance dosage
Presence of urinary lithiasis | Through study completion, an average of 1 year
  Serum creatinine and clearance dosage
Presence of cardiovascular complications | Through study completion, an average of 1 year
  Defined as ischemic cardiopathy

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU Angers, Angers
  - Centre Hospitalier Le Mans, Le Mans
  - CHU Limoges, Limoges
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - AP-HP La Pitié Salpétrière, Paris

IPD SHARING:
Plan to Share IPD: Undecided